CLINICAL TRIAL: NCT01184651
Title: "Gender Development in Early Adolescence: Prenatal Hormones and Family Socialization"
Brief Title: Tweens to Teens Project at Penn State
Acronym: T2T@PSU
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sheri Berenbaum, Professor of Psychology and Pediatrics, Penn State University
Other Study IDs: PSU ORP#30695; 1R01HD057930-01A1 (NIH)
Record Dates: First submitted 2010-08-02; First posted 2010-08-19 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Congenital Adrenal Hyperplasia; CAH; sex differences; adolescence; androgen; behavior; gender development
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Behavior | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples of saliva will be collected from participants with CAH for genetic testing (specific mutations of CYP21 gene) and to obtain hormone levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Girls: Girls with 21-hydroxylase deficiency (21-OHD) congenital adrenal hyperplasia (CAH) ages 10-13
  Interventions: Behavioral: Questionnaires/Interviews
- Parents: Parent, guardian, or significant caretaker of girls with CAH
  Interventions: Behavioral: Questionnaires/Interviews

INTERVENTIONS:
Behavioral: Questionnaires/Interviews — Girls answer questions about activities and interests, school, feelings about being a girl, stage of physical development, and family relationships during a home interview , provide saliva samples, and participate in phone interviews to answer questions about daily activities .
  Groups: Girls
Behavioral: Questionnaires/Interviews — Parents complete questionnaires about their daughter's activities, interests, and behaviors, educational goals, family demographics and relationships, grades, diagnosis and treatment of her CAH, their own activities, interests, and thoughts and feelings about being male or female. Parents answer questions during phone interviews about their daughters daily activities.
  Groups: Parents

SUMMARY:
The goal of this study is to help investigators to understand more about the development of characteristics related to being male or female (what is called gender development). The investigators will study girls with congenital adrenal hyperplasia (CAH) aged 10 to 13 to learn more about the girls' interests and activities, thoughts and feeling about being female, and family relationships. This will help investigators to understand the ways in which gender development is shaped by hormones and family relationships.

DETAILED DESCRIPTION:
Interviewers will visit girls in their home when it is convenient for the family. Girls will answer questions about the things they do and are interested in, how they think and feel, and complete some cognitive tasks. Girls will also provide saliva so we can examine their hormones and determine the CAH gene mutation they have. Parents will also be asked to complete questionnaires about their own activities and interests and about their daughter's behavior.

Shortly after the home visit, interviewers will telephone girls and their parents on several days and ask what the girls did during the day.

ELIGIBILITY:
Inclusion Criteria:

* Girls with classical or non-classical CAH due to 21-OHD
* Girls will be aged 10-13 years at initial recruitment
* Parents will include biological mothers and fathers as well as step-parents and/or other guardians/significant caregivers
* Parents/guardians may range in age from 18 years of age to 65 years of age.

Exclusion Criteria:

* Girls who are not within the age range of 10-13 years old at initial recruitment
* CAH not due to the 21-OHD form

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will study girls with the 21-hydroxylase deficiency (21-OHD) form of congenital adrenal hyperplasia (CAH) aged 10 to 13. Parents of participants are also included.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2009-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheri A Berenbaum, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, Dept. of Psychology - Tweens to Teens Project, University Park, Pennsylvania, United States